CLINICAL TRIAL: NCT03074916
Title: Outcomes of Motion-preserving Surgery and Arthrodesis at the Distal Interphalangeal (DIP) Joint
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: DIP_Silicone_retro
Record Dates: First submitted 2017-02-23; First posted 2017-03-09 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Distal Interphalangeal Arthroplasty; Distal Interphalangeal Arthrodesis
MeSH Terms: interventions — Arthrodesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DIP arthroplasty
  Interventions: Device: DIP arthroplasty or arthrodesis
- DIP arthrodesis
  Interventions: Device: DIP arthroplasty or arthrodesis

INTERVENTIONS:
Device: DIP arthroplasty or arthrodesis — Arthroplasty of the DIP Joint or arthrodesis of the DIP joint

SUMMARY:
The objective of this project is to investigate the subjective and clinical outcome in patients at least one year after DIP arthroplasty and compare them to matched patients with an arthrodesis.

The primary endpoint is the satisfaction with the treatment result of in the motion-preserving DIP surgery at follow-up.

ELIGIBILITY:
Inclusion Criteria:

Arthroplasty group:

* DIP silicone arthroplasty at least one year ago
* Informed consent as documented by signature

Arthrodesis group:

* Matched patients with an DIP arthrodesis
* Informed consent as documented by signature

Exclusion Criteria:

Arthroplasty group:

* Silicone arthroplasty at the thumb IP joint
* Major surgery at another joint (PIP arthroplasty, thumb trapeziectomy) less than 6 months ago
* Legal incompetence
* German language barrier to complete the questionnaires

Arthrodesis group:

* Arthroplasty at another DIP joint
* Major surgery at another joint (PIP arthroplasty, thumb trapeziectomy) less than 6 months ago
* Legal incompetence
* German language barrier to complete the questionnaires

Ages: 18 Years to 111 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a DIP arthroplasty at least one year ago Matched patients with a DIP arthrodesis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
satisfaction with the treatment result of the motion-preserving DIP surgery at follow-up | at least 1 year up to 7 years
  Question to be answered on a 5 Point Likert scale

SECONDARY OUTCOMES:
Michigan Hand Questionnaire | at least 1 year up to 7 years
  Questionnaire about Hand function scored 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No